CLINICAL TRIAL: NCT03420209
Title: The Effect of Proprioceptive Neuromuscular Facilitation Technique on Respiratory Functions, Functional Capacity, Muscle Force, Posture, Activity of Daily Living, Quality of Life for Children With Chronic Pulmonary Diseases.
Brief Title: The Effect of Proprioceptive Neuromuscular Facilitation (PNF) Technique for Children With Chronic Pulmonary Diseases.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Gamze Baskent, Pincipal İnvestigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1493
Record Dates: First submitted 2018-01-27; First posted 2018-02-05 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Chronic Respiratory Disease; Cystic Fibrosis; Bronchiectasis
Keywords: proprioceptive neuromuscular facilitation; respiratory functions; elastic band; posture
MeSH Terms: conditions — Cystic Fibrosis; Bronchiectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group applying PNF technique (Experimental): The experimental goup who are applying PNF technique with elastic bands for the upper extremities. Before the group will perform stretching and resisted exercises at the warming up period, after they will do PNF exercises with elastic bands on two PNF pattern for the upper extremities and finally they will do some stretching exercises for the cool down period. The programme will continue for 30-45 minutes, three times a week, for 12 weeks. They will work one by one with a physical therapist.
  Interventions: Behavioral: Group applying PNF technique
- Home Programme (No Intervention): This group will perform only breathing exercises daily at home during 12 weeks.

INTERVENTIONS:
Behavioral: Group applying PNF technique
  Arms: Group applying PNF technique

SUMMARY:
Cystic fibrosis and bronchiectasis are the most seen problems in children with chronic pulmonary diseases. İt is a genetic, chronic system disease that reduces life expectancy, and life quality as well. Chronic lung disease , malnutrition, and reduced activity, caused by disease lead to postural disorders. Muscle force, endurance, activity of Daily living are adversely affected. İn the treatment pulmonary rehabilitation are using. Airway clearance technique, pulmonary exercises, upper extremity ergometer, dumbbells, elastic bands, proprioceptive neuromuscular facilitation technique are applying. Resistance training using elastic bands has become an increasingly common intervention aiming to improve function by increasing muscular strength. İn one study indicated that muscle strength can be improved through three dimensional spiral large scale resistive exercises using proprioceptive neuromuscular facilitation. İn the literature there isn't any research , uses elastic bands with proprioceptive neuromuscular facilitation for the upper extremity and evaluating pulmonary functions, posture, quality of life, muscle force.

The aim of this study is giving exercises programme with proprioceptive neuromuscular facilitation and elastic bands and to evaluate pulmonary muscle force, pulmonary functions, posture, activity of daily living, quality of life, functional capacity. And to evaluate the effect of treatment programme on these parameters.

The subjects were divided in two groups. An experimental group three times a week for 12 weeks will perform proprioceptive neuromuscular facilitation exercises with elastic bands, and pulmonary exercises. The control group will apply only pulmonary exercises at home programme.

DETAILED DESCRIPTION:
Participants: All participants with chronic respiratory disease were recruited from a Istanbul University Medical Faculty, Allergy Department. All treatments were performed in the same hospital.

Sample Size: Sample size was calculated with power analysis. Pass 11 Home programme was used. α=0,05, β=0,6, 1- β=0,94 was determined. İf Sample size was defined 20 experimental and 20 control group the power obtained %95. Using two-sided two sample t-test with alpha 0,05 standard deviations were 5,0 and 4,0.

Procedure: Forty chronic respiratory disease patient were assessed between the age of 10-18 years old. The patients were found to be suitable for inclusion criteria of the study.Randomisation was performed by using randomisation function of Microsoft Office Excel programme by another researcher (ARO). Random number generator of Microsoft Office Excel Software gave a random number between 0 and 1 to the each treatment columns which were created by ARO. Sorting the random number row from the largest to the smallest number was performed by the sort and filter menu.After the randomisation,assessments at baseline and the patients were divided two groups. The experimental group was treated one by one with one physical therapist three times a week during a session for 30-45 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 10-18 years
2. Walking alone
3. The children with chronic pulmonary diseases who can cooperate
4. Children who can accommodate to the programme
5. The family who gave informed consent
6. The children who are didn't at the acute exacerbation attack.

Exclusion Criteria:

1. The children can't walk alone
2. The children with chronic pulmonary diseases who can't cooperate
3. The family who didn't gave informed consent
4. The children who are at the acute exacerbation attack.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary function test | 12 weeks
  This test evaluates respiratory functions. Dynamic pulmonary volumes will evaluate.

SECONDARY OUTCOMES:
Posture Analysis | 12 weeks
  Plonk image measurement system is a posture analysis method evaluated on the computer software programme. We place the markers on the anatomic points of the body. We take a Picture with the camera. There is a 3 meter distance with the camera and the child. We take a Picture three times on the sagittal, frontal and lateral side.
6 Minutes Walk Test | 12 weeks
  This test was used to evaluate functional capacity. They are walking during six minutes on the corridor of 30 m. İf there is a fatigue they can have a rest. And they can continue to walk. We have to measure the distance of walking during six minutes. Before and after the test we have to measure the dyspnea and level of fatigue with perceived exertion scale.
6 Minutes Pegboard and Ring Test | 12 weeks
  İt measures functional capacity on the upper extremities of the body. Briefly, subjects were asked to move as many rings (each ring weighed 50 g; Zhan et al had used rings weighing half an ounce) as possible in 6 minutes, and the score was the number of rings moved during the 6-minute period. Pulse oxygen saturation was measured during the test. Scores for dyspnea were evaluated using a modified perceived exertion scale (0-10)13 immediately after the test.
The Pediatric Quality of Life Inventory (PedsQ-L)test | 12 weeks
  This was used to measure quality of life for children. There are subgroups measuring physically, social, sensory and the problems living at school.
Muscle testing | 12 weeks
  Muscle testing with the hand held dynamometer. Upper extremity muscle force will evaluate with the dynamometer.
Maximal inspiratory pressure and Maximal expiratory pressure measurement | 12 weeks
  Maximal inspiratory pressure and Maximal expiratory pressure will measure the respiratory muscle force with the Micro respiratory pressure measure.
Glitter-Activity of Daily Living test, Activity of Daily living measurement | 12 weeks
  In this test the patient reports the activities that promote discomfort during daily living activities. During its execution, functional capacity is evaluated by the time spent to perform a circuit that consists of global activities as walking, climbing up-and-down stairs, and trunk and upper limbs movements. The lower time spent the better is the functional condition. This test will measure functional capacity and easy to use.

CONTACTS AND LOCATIONS:
Overall Officials: Zerrin Dr Yigit, Prof, Study Director — Istanbul University, Cardiology Institute, Cardiology Department
Locations (1):
- Gamze Baskent, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mays RJ, Goss FL, Nagle EF, Gallagher M Jr, Haile L, Schafer MA, Kim KH, Robertson RJ. Cross-validation of Peak Oxygen Consumption Prediction Models From OMNI Perceived Exertion. Int J Sports Med. 2016 Sep;37(10):831-7. doi: 10.1055/s-0042-103029. Epub 2016 Jul 13. PMID 27410768
- [Result] Bass JL, Corwin M, Gozal D, Moore C, Nishida H, Parker S, Schonwald A, Wilker RE, Stehle S, Kinane TB. The effect of chronic or intermittent hypoxia on cognition in childhood: a review of the evidence. Pediatrics. 2004 Sep;114(3):805-16. doi: 10.1542/peds.2004-0227. PMID 15342857
- [Result] Kamel TB, Abd Elmonaem MT, Khalil LH, Goda MH, Sanyelbhaa H, Ramzy MA. Children with chronic lung diseases have cognitive dysfunction as assessed by event-related potential (auditory P300) and Stanford-Binet IQ (SB-IV) test. Eur Arch Otorhinolaryngol. 2016 Oct;273(10):3413-20. doi: 10.1007/s00405-016-4044-z. Epub 2016 Apr 13. PMID 27075686
- [Result] Rossi UG, Owens CM. The radiology of chronic lung disease in children. Arch Dis Child. 2005 Jun;90(6):601-7. doi: 10.1136/adc.2004.051383. PMID 15908625
- [Result] Arikan H, Yatar I, Calik-Kutukcu E, Aribas Z, Saglam M, Vardar-Yagli N, Savci S, Inal-Ince D, Ozcelik U, Kiper N. A comparison of respiratory and peripheral muscle strength, functional exercise capacity, activities of daily living and physical fitness in patients with cystic fibrosis and healthy subjects. Res Dev Disabil. 2015 Oct-Nov;45-46:147-56. doi: 10.1016/j.ridd.2015.07.020. Epub 2015 Aug 1. PMID 26241869
- [Result] Santana-Sosa E, Gonzalez-Saiz L, Groeneveld IF, Villa-Asensi JR, Barrio Gomez de Aguero MI, Fleck SJ, Lopez-Mojares LM, Perez M, Lucia A. Benefits of combining inspiratory muscle with 'whole muscle' training in children with cystic fibrosis: a randomised controlled trial. Br J Sports Med. 2014 Oct;48(20):1513-7. doi: 10.1136/bjsports-2012-091892. Epub 2013 May 16. PMID 23681502
- [Result] Alison JA, Regnis JA, Donnelly PM, Adams RD, Sutton JR, Bye PT. Evaluation of supported upper limb exercise capacity in patients with cystic fibrosis. Am J Respir Crit Care Med. 1997 Nov;156(5):1541-8. doi: 10.1164/ajrccm.156.5.97-02034. PMID 9372673
- [Result] Wells GD, Wilkes DL, Schneiderman JE, Thompson S, Coates AL, Ratjen F. Physiological correlates of pulmonary function in children with cystic fibrosis. Pediatr Pulmonol. 2014 Sep;49(9):878-84. doi: 10.1002/ppul.22928. Epub 2013 Oct 25. PMID 24166871
- [Result] Sharman MJ, Cresswell AG, Riek S. Proprioceptive neuromuscular facilitation stretching : mechanisms and clinical implications. Sports Med. 2006;36(11):929-39. doi: 10.2165/00007256-200636110-00002. PMID 17052131
- [Result] Williams JG, Odley JL, Callaghan M. Motor Imagery Boosts Proprioceptive Neuromuscular Facilitation in the Attainment and Retention of Range-of -Motion at the Hip Joint. J Sports Sci Med. 2004 Sep 1;3(3):160-6. eCollection 2004 Sep. PMID 24482593
- [Result] Porto EF, Castro AA, Nascimento O, Oliveira RC, Cardoso F, Jardim JR. Modulation of operational lung volumes with the use of salbutamol in COPD patients accomplishing upper limbs exercise tests. Respir Med. 2009 Feb;103(2):251-7. doi: 10.1016/j.rmed.2008.08.018. Epub 2008 Oct 19. PMID 18930646
- [Result] Seo K, Cho M. The effects on the pulmonary function of normal adults proprioceptive neuromuscular facilitation respiration pattern exercise. J Phys Ther Sci. 2014 Oct;26(10):1579-82. doi: 10.1589/jpts.26.1579. Epub 2014 Oct 28. PMID 25364117
- [Result] Areas GP, Borghi-Silva A, Lobato AN, Silva AA, Freire RC Jr, Areas FZ. Effect of upper extremity proprioceptive neuromuscular facilitation combined with elastic resistance bands on respiratory muscle strength: a randomized controlled trial. Braz J Phys Ther. 2013 Nov-Dec;17(6):541-6. doi: 10.1590/S1413-35552012005000131. Epub 2013 Nov 1. PMID 24346292
- [Result] Colado JC, Pedrosa FM, Juesas A, Gargallo P, Carrasco JJ, Flandez J, Chupel MU, Teixeira AM, Naclerio F. Concurrent validation of the OMNI-Resistance Exercise Scale of perceived exertion with elastic bands in the elderly. Exp Gerontol. 2018 Mar;103:11-16. doi: 10.1016/j.exger.2017.12.009. Epub 2017 Dec 17. PMID 29262307